CLINICAL TRIAL: NCT05129306
Title: Impact of RYALTRIS® (Olopatadine Hydrochloride / Mometasone Furoate Monohydrate) Nasal Spray on Patients' Reported Outcomes
Brief Title: Impact of RYALTRIS® Nasal Spray on Patients' Reported Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty recruiting participants with current strategy
Sponsor: Community and Patient Preference Research Pty Ltd (Industry)
Collaborators: Seqirus Limited (Unknown); Glenmark Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20210902_1
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis
Keywords: Patient outcomes; Patient satisfaction; Quality of Life
MeSH Terms: conditions — Rhinitis, Allergic; Patient Satisfaction | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with moderate to severe Allergic Rhinitis who have been prescribed RYALTRIS® nasal spray by their healthcare professional. Observational.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — In this observational study, participants with moderate to severe Allergic Rhinitis who were initiated on Ryaltris® nasal spray by their healthcare professional will complete an online survey before commencement of treatment and then at days 1, 7, and 14 from treatment initiation. Survey completion at day 28 after treatment initiation will be optional for participants based on ongoing use of RYALTRIS®.

SUMMARY:
A real world evidence study that aims to understand the impact of RYALTRIS® nasal spray in patients with Allergic Rhinitis over a 28-day period.

DETAILED DESCRIPTION:
The aim of this research is to develop a greater understanding of satisfaction with RYALTRIS® nasal spray in patients with Allergic Rhinitis (AR). There is currently no real-world evidence for patient satisfaction data with RYALTRIS® nasal spray. To address this knowledge gap and add to clinically relevant data to support Quality of Life (QoL) and patient reported outcomes, this research will evaluate the impact on quality of life (symptom control), using a Visual Analogue Scale (VAS), following initiation of RYALTRIS® to explore the relationship between baseline and subsequent QoL scores among patients initiated on RYALTRIS®.

ELIGIBILITY:
Inclusion Criteria:

AR patients (moderate-to-severe SAR or PAR) with or without conjunctivitis who meet the following criteria will be offered the opportunity to participate in the study:

* Patients above 18 years old
* Fluent in English
* Patients newly prescribed RYALTRIS® who have not yet initiated treatment
* Willing and able to provide consent to participate

Exclusion Criteria:

Potential participants will be excluded if they:

* Are employed by a pharmaceutical company (to avoid conflict of interest)
* Are employed by a vaccine company (to avoid conflict of interest)
* Do not have access to the internet (to ensure validity of the data)
* Are unable to read and understand English (to ensure validity of the data)
* are currently or have previously been on RYALTRIS®

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The primary population will be patients with moderate to severe Seasonal Allergic Rhinitis (SAR) or Perennial Allergic Rhinitis (PAR) in Australia who have been newly prescribed RYALTRIS® for management of their disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 28 days
  The primary study endpoint is the overall VAS score to determine improvement of Allergic Rhinitis symptoms and quality of life.

SECONDARY OUTCOMES:
Overall Allergic Rhinitis nasal symptoms | 28 days
  Response to a visual analogue scale about their Allergic Rhinitis nasal symptoms
Overall Allergic Rhinitis ocular symptoms | 28 days
  Response to a visual analogue scale about their Allergic Rhinitis ocular symptoms
Sleep quality | 28 days
  Response to a visual analogue scale about their sleep quality
Daily outdoor activities | 28 days
  Response to a visual analogue scale about their daily outdoor activities
Work productivity | 28 days
  Response to a visual analogue scale about their work productivity

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fifer, PhD, Principal Investigator — Community and Patient Preference Research Pty Ltd
Locations (1):
- Community and Patient Preference Research Pty Ltd, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Australian Institute of Health and Welfare 2019. Allergic rhinitis ('hay fever'). Cat. no. PHE 257. Canberra: AIHW. Viewed 01 May 2020, https://www.aihw.gov.au/reports/chronic-respiratory-conditions/allergic-rhinitis-hay-fever/contents/allergic-rhinitis
- [Background] Meltzer EO, Garadi R, Laforce C, Chadwick SJ, Berger WE, Gross G, Edwards MR, Crenshaw K, Wall GM. Comparative study of sensory attributes of two antihistamine nasal sprays: olopatadine 0.6% and azelastine 0.1%. Allergy Asthma Proc. 2008 Nov-Dec;29(6):659-68. doi: 10.2500/aap.2008.29.3181. Epub 2008 Dec 6. PMID 19144261
- [Background] Meltzer EO, Hadley J, Blaiss M, Benninger M, Kimel M, Kleinman L, Dupclay L, Garcia J, Leahy M, Georges G. Development of questionnaires to measure patient preferences for intranasal corticosteroids in patients with allergic rhinitis. Otolaryngol Head Neck Surg. 2005 Feb;132(2):197-207. doi: 10.1016/j.otohns.2004.10.010. PMID 15692526
- [Background] Price D, Klimek L, Galffy G, Emmeluth M, Koltun A, Kopietz F, Nguyen DT, van Weissenbruch R, Pohl W, Kuhl HC, Scadding G, Mullol J. Allergic rhinitis and asthma symptoms in a real-life study of MP-AzeFlu to treat multimorbid allergic rhinitis and asthma. Clin Mol Allergy. 2020 Aug 6;18:15. doi: 10.1186/s12948-020-00130-9. eCollection 2020. PMID 32782442